CLINICAL TRIAL: NCT00831883
Title: Partner-Specific HIV Risk Reduction Intervention for Drug-Using Incarcerated Adolescents
Brief Title: Partner-Specific HIV Risk Reduction Intervention for Drug-Using Adolescents
Acronym: GET UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Collaborators: University of Rhode Island (Other)
Responsible Party: Principal Investigator, Cynthia Rosengard, Cynthia Rosengard, Ph.D., Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 08-0128; R01DA022921-03 (NIH)
Record Dates: First submitted 2009-01-28; First posted 2009-01-29 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Sexually Transmitted Diseases; Substance-Related Disorders
Keywords: Adolescent; Adolescent behavior; Health behavior; Sexual Behavior; Incarceration; Behavioral Intervention; Risk Reduction Behavior
MeSH Terms: conditions — Sexually Transmitted Diseases; Substance-Related Disorders; Adolescent Behavior; Health Behavior; Sexual Behavior; Risk Reduction Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Partner Specific IMB (Experimental): partner-specific HIV risk reduction intervention
  Interventions: Behavioral: Partner-Specific IMB-based HIV risk reduction intervention
- HLS (Placebo Comparator): 5 session psychoeducational group, designed to provide equivalent time and attention, that focuses on the importance of maintaining a good diet, exercise, and developing health skills.
  Interventions: Behavioral: Healthy Lifestyle

INTERVENTIONS:
Behavioral: Partner-Specific IMB-based HIV risk reduction intervention — 5 session partner-specific HIV risk reduction group intervention based on the Information-Motivation-Behavioral Skills model.
  Arms: Partner Specific IMB
Behavioral: Healthy Lifestyle — 5 session psychoeducational group, designed to provide equivalent time and attention, that focuses on the importance of maintaining a good diet, exercise, and developing health skills.
  Arms: HLS

SUMMARY:
The purpose of this study is to develop and pilot test a partner-specific HIV risk reduction intervention for currently or recently incarcerated adolescents who report problematic substance use.

DETAILED DESCRIPTION:
Incarcerated adolescents represent a group at high risk for health consequences associated with risky sexual behaviors. Condom use is more common with non-main than main sex partners and substance use in conjunction with sexual risk also appears to vary by partner type. The research team will conduct a small randomized trial to pilot test a partner-specific HIV risk reduction intervention for currently or recently incarcerated adolescents who report problematic substance use. Participants will be randomized to a 5 session HIV risk reduction group intervention based on the Information-Motivation-Behavioral Skills model, or a 5 session healthy lifestyles psychoeducation intervention, and then reassessed 3 months after their access to the general community is reinstated. The main hypothesis is that participants in the HIV risk reduction intervention condition will have lower levels of sex-related HIV risk behavior and of substance use in conjunction with sexual risk, relative to those in a healthy lifestyles psychoeducation intervention.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking ability
* unprotected vaginal, anal, or oral intercourse at least once in the 6 months prior to incarceration or placement
* marijuana use disorders, other non-injection drug use disorders, or substance use by a sexual partner during a sexual episode in the six months prior to incarceration or placement
* sentence or placement length between 2 and 12 months
* must plan to remain in the area for the 6 months following their release from the facility
* must be willing to provide two pieces of contact information for follow-up

Exclusion Criteria:

* signs of psychosis (assessed through clinical assessment)

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 59 (Actual)
Dates: Start 2009-02; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
lower levels of sex-related HIV risk behavior | 3 months

SECONDARY OUTCOMES:
knowledge about STI transmission | 3 months
partner-specific perceptions of STI risks | 3 months
social norms, expectations and personal attitudes regarding partner-specific sexual behavior | 3 months
partner-specific behavioral and communication skills | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Rosengard, PhD, MPH, Principal Investigator — Women & Infants of Rhode Island
Locations (1):
- Women & Infants Hospital of Rhode Island, Providence, Rhode Island, United States